CLINICAL TRIAL: NCT06002074
Title: Impact of the Stress Management and Resilience Training (SMART) Program on Quality of Life in Patients with Inflammatory Bowel Diseases
Brief Title: SMART Program Impact on Quality of Life in Inflammatory Bowel Diseases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Decision to end study
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Victor Chedid, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-004024
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Diseases; Stress
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stress management and resilience training (Experimental): Subjects will receive a 1.5 hour one-on-one stress management and resilience consult by a certified SMART trainer followed by 16 week self-guided on-line training.
  Interventions: Behavioral: Stress Management and Resilience Training Program

INTERVENTIONS:
Behavioral: Stress Management and Resilience Training Program — One-on-one stress management and resilience consultation by a certified SMART trainer followed by self-guided on-line training consisting of 4 modules.
  Other Names: SMART

SUMMARY:
This research study is being done to look at the impact of a Stress Management and Resilience Training (SMART) Program on the quality of life and healthcare utilization of patients with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* History of IBD defined by a physician global assessment (PGA) of quiescent, mild, moderate, or severe disease.
* Access to internet/device such as smart phone, tablet, or computer
* Patient reports stress as a trigger to their GI symptoms

Exclusion Criteria:

* Corticosteroids in the previous 3 months
* Elicit substance use (including medical marijuana)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Change in Inflammatory Bowel Disease (IBD) Quality of Life (QOL) | Baseline, approximately 20 weeks
  Measured by self-reported 32-item Quality of Life in Inflammatory Bowel Disease Questionnaire (IBDQ) designed to assess feelings about symptoms as a results of IBD over the last 2 weeks. Responses to each question are scored on a 7-point Likert scale ranging from 1 (a very severe problem) to 7 (not a problem). Possible total scores range from 32 to 224, where higher scores indicate better outcome/better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Victor G. Chedid, M.D., M.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No